CLINICAL TRIAL: NCT02550600
Title: EXODUS: Extracorporeal Lung Assist Device in Acute Lung Impairment: A Randomized Controlled Study
Brief Title: Extracorporeal Lung Assist Device in Acute Lung Impairment
Acronym: EXODUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Novalung GmbH, Heilbronn, Germany (Unknown); Studiensekretariat Intensivmedizin; II. Medizinische Klinik; Klinikum rechts der Isar; Munich (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXO_1
Record Dates: First submitted 2015-07-24; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Acute lung impairment; Extracorporeal lung assist; ECMO; ECLA; Murray-score; SOFA-score
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention: iLA activve treatment. iLA activve treatment also requires anticoagulation with un-fractionized heparin and pre-defined PTT-goals (45s-60s depending on blood flow).
  Interventions: Procedure: iLA activve treatment
- Control group (Active Comparator): Controls: standard care according to good clinical practice and recent guidelines; no extracorporeal lung assist.
  For ethical reasons patients of the control group can be treated with iLA activve after fulfilling the primary endpoint criterium of an increase in SOFA ≥3 points. These cross-over patients will be analyzed as controls ("intention to treat").
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: iLA activve treatment — iLA activve is aimed at efficient extracorporeal membrane oxygenation with an initial blood flow of ≥2L/min. The length of therapy is at the discretion of the treating physician.
  Treating physicians are recommended to use a pre-specified algorithm to optimize the extracorporeal lung assist (choice of cannulas and oxygenator, titration of blood flow and sweep gas flow). Primary/mandatory goals are pO2≥65mmHg, P_peak ≤30cm H2O, TV ≤6ml/kg PBW and pH ≥7.25. Secondary suggested goals are setting the PEEP level within the limits suggested by the ARDSnet low and high PEEP strategy, 35mmHg ≤ pCO2 ≤45mmHg, Delta-pressure (= P_peak - PEEP) ≤15 cm H2O and P_peak ≤25 cm H2O.
  iLA activve treatment also requires anticoagulation with un-fractionized heparin (PTT-goal 45s-60s depending on blood flow).
  Other Names: ECMO; Extra-corporeal lung assist
  Arms: Intervention group
Procedure: Control group — The controls will be treated according to the recent guideline of the German Sepsis Society and the German Interdisciplinary Association of Intensive Care and Emergency Medicine and good clinical practice including lung-protective ventilation with low tidal volume (LTV), moderate hypercapnia, PEEP according to ARDSnet, adjunctive measures (e.g. prone positioning; neuromuscular blockers as appropriate) and treatment of the underlying disease as applied in the experimental group.
  There will be no sham treatment of iLA activve.in the controls. All adjunctive measures (e.g. prone positioning; neuromuscular blockers as appropriate) are also available for the intervention group.
  Arms: Control group

SUMMARY:
The purpose of this study is to compare the effect of interventional Lung Assist iLA activve to standard therapy in mechanically ventilated patients with severe acute lung impairment. Hypothesis: iLA(active) reduces the incidence of an increase in SOFA-Score of ≥3 points (or death) within 28 days compared to standard treatment.

DETAILED DESCRIPTION:
Background:

Mechanical ventilation in patients with acute lung impairment further injures the lungs by inspiration forces and inflammatory response. Large efforts have been invested in reducing ventilator-associated lung damage by lower tidal volumes. However, benefits are limited by potential harms of permissive hypercapnia.

Therefore, extracorporeal membrane oxygenation (ECMO) and CO2-removal have been studied for more than 40 years. However, ECMO remained restricted to few specialized centres capable to provide extensive resources. Transfer of patients implicates loss of time and risks of transportation. Therefore, less invasive devices have been developed, including "pump-less "extracorporeal lung assist" (pECLA) and pump-driven ECLA (e.g. iLA activve). Despite pilot trials supporting feasibility, safety and efficient oxygenation and decarboxylation by pump-driven ECLA, there are no randomized controlled trials (RCT) proving a benefit regarding long-term endpoints.

Objectives:

Therefore, the aim of this multicentre RCT is to compare the outcome of 150 patients with early (after ≤96h of mechanical ventilation) acute lung impairment treated by pump-driven ECLA with iLA activve with a blood flow of at least 1L/min vs. 150 controls with standard intensive care including low tidal volume ventilation.

Main inclusion and exclusion criteria:

While most trials on ECMO and (p)ECLA included patients in a rescue scenario with severe and persisting ARDS, earlier inclusion also implicates modified inclusion criteria: A cumulative Murray score of ≥6 points without radiological points is the most important inclusion criterion. At least four points must result from pO2/FiO2 (mandatory pO2/FiO2<300mmHg) and PEEP criteria of the Murray score. In order to provide sufficient time for conservative attempts to optimize ventilation, inclusion criteria can be fulfilled for a maximum of 48h before inclusion as long as the patient can be included within a maximum of 96h of mechanical ventilation.

Primary efficacy endpoint:

Incidence of an increase in SOFA-Score ≥3 points or death within 28 days.

Statistical analyses:

Generalized linear mixed model (logit link function) will be used to compare the primary efficacy endpoint, the proportion of patients with an increase in SOFA of ≥3 points or death within 28d, between the two groups. In this analysis the random factor variable study centre and anticoagulation therapy will be considered as adjustment variables. The test of group effect estimated by the multivariable mixed logistic model will be conducted at a two-sided 0.05 level of significance.

The primary efficacy analysis will be based on the intention-to-treat population. Missing values of SOFA score will be replaced by last-value carry forward approach.

Survival status of lost to follow-up patients will be replaced conservatively: missing survival status will be replaced by attribute "death" for patients in the verum arm and replaced by attribute "alive" for patients in the standard treatment arm.

A supportive complete case and per-protocol analysis will be conducted for purpose of sensitivity analysis of the primary endpoint. Further sensitivity analyses will be provided to evaluate robustness of results in regard to unexpected circumstances (e.g. impact of 'cross-over' patients who are not treated as randomized but are required to be analyzed as randomized (ITT-principle)). Secondary endpoints will be analyzed in an exploratory manner.

Chi-Square test or Fisher-exact test will be used to compare categorical data. For comparisons of continuous data between groups non-parametric tests (Kruskal-Wallis test, Mann-Whitney-U test) will be performed. 95% confidence intervals will be calculated for relevant measurements. SAS software (version 4.9 or future follow-up version).

ELIGIBILITY:
Inclusion Criteria:

* Potentially reversible lung failure AND
* Cumulative Murray score ≥6 points without radiological points for a maximum of 48h AND
* Cumulative Murray score ≥4 points for pO2/FiO and PEEP AND
* Cumulative Murray score ≥1 point for pO2/FiO
* Mechanical ventilation for ≤96h AND
* Age ≥ 18 years.

Exclusion Criteria:

* SOFA-Score >20
* Life expectancy <24h
* mechanical ventilation >96h
* Heparin-induced thrombopenia
* Intracranial bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of an increase in SOFA-Score ≥3 points or death within 28 days | 28 days

SECONDARY OUTCOMES:
Death or severe disability after 6 months defined as confinement to bed and inability to wash or dress alone | 6 months
Mortality | 28 days, 60 days, ICU-stay
Ventilator free days | 28 days, ICU stay
Single organ failures as assessed by SOFA | 28 days, ICU stay
Prediction of outcome (Primary endpoint: Incidence of an increase in SOFA-Score ≥3 points or death within 28 days) | 28 days
  Uni- and multivariate analysis of the predictive capabilities of baseline values of extravascular lung water index and graduation of ARDS (AECC- and Berlin definition of ARDS, Murray-score)
Safety analysis assessed by documentation of complications and side effects potentially related to iLA activve and/or conventional therapy including complications associated to cannulation and extracorporeal circuit, | 6 months
  thrombosis, pulmonary embolism, pneumothorax, use of tube thoracostomies
Meta-analysis | 6 months
  Meta-analysis of this study and other high-quality RCTs on extracorporeal lung Support regarding survival to 6 months without disability, all cause mortality on day 60.
Resource use and economic outcomes | 6 months
  Comparison of resource use based on DRG-calculation
Early vs. late intervention | 6 months
  Comparison of outcome of patients with early iLA activve (Intervention group) to late iLA activve (Control group with cross-over): survival to 6 months without disability, mortality after 28 days, 60 days and 6 months.
Prediction of outcome (Death or severe disability after 6 months defined as confinement to bed and inability to wash or dress alone) | 6 months
  Uni- and multivariate analysis of the predictive capabilities of baseline values of extravascular lung water index and graduation of ARDS (AECC- and Berlin definition of ARDS, Murray-score)
Association of the fluid balance to the primary endpoint (Incidence of an increase in SOFA-Score ≥3 points or death within 28 days) | 28 days
  Uni- and multivariate analysis regarding the association of the cumulative fluid balance with the primary endpoint
Association of the fluid balance to the secondary endpoint "death or severe disability after 6 months defined as confinement to bed and inability to wash or dress alone)" | 6 months
  Uni- and multivariate analysis regarding the association of the cumulative fluid balance with the secondary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber, MD, Principal Investigator — II. Medizinische Klinik; Klinikum rechts der Isar; Ismaningerstrasse 22; D-81675 München; Germany
Locations (8):
- Medical University of Vienna/General Hospital of Vienna, Vienna, Austria
- Germany (5):
  - Klinik für Intensivmedizin; Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Abteilung für Intensivmedizin; Krankenhaus Barmherzige Brüder; München, Munich
  - I. Medizinische Klinik; Klinikum rechts der Isar; Technische Universität München, Munich
  - II. Medizinische Klinik; Klinikum rechts der Isar; Technische Universität München, München
  - Klinik für Anästhesiologie; Klinikum rechts der Isar; Technische Universität München, München
- Department of Anaesthesiology and Intensive Therapy; University of Szeged, Szeged, Hungary
- St. Bartholomew's & London Chest Hospitals, London, United Kingdom